CLINICAL TRIAL: NCT04296084
Title: Determination of Upper Extremity Kinematics During Walking in Healthy Individuals
Brief Title: Upper Extremity Kinematics During Walking
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Güngör Beyza ÖZVAR, MSc physiotherapist, Hacettepe University
Other Study IDs: Kinematic analysis in walking
Record Dates: First submitted 2020-02-27; First posted 2020-03-05 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-05

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy individuals: Volunteer healthy individuals who are between the ages of 20-40 and who do not have any medical condition to affect gait or arm swing.

SUMMARY:
Our aim is to investigate the upper extremity kinematics during walking in healthy individuals.

DETAILED DESCRIPTION:
Determination of Upper Extremity Kinematics During Walking

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20 and 40 years individuals
* Without any medical condition that would affect gait or arm swing

Exclusion Criteria:

* People with upper or lower limb asymmetry

Ages: 20 Years to 40 Years | Sex: All
Age Groups: Adult
Study Population: Healthy individuals in the age of 20-40 years
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-05-10 (Actual); Study Completion 2020-05-12 (Actual)

PRIMARY OUTCOMES:
Kinematic analysis | up to 20 weeks
  For kinematic analysis, MVN BIOMECH Awinda MTW2-3A7G6 sensors (Xsens Technologies B.V. Enschede, The Netherlands) were used. A Kalman filter (Xsens Kalman Filter, XKF) was used for 3D reconstruction of body segment position and orientation. IMU sensors were placed in accordance with the anatomical regions found in the directive issued by the International Biomechanics Association. Joint kinematic data of bilateral upper limb, lower limb and trunk were recorded with IMU sensors and wireless station. Xsens MVN Studio 4.6 was used to track IMU orientations according to the world-based coordinate framework. To make an effective analysis, gloves, vests and velcro were used to attach sensors to the extremities and body.

SECONDARY OUTCOMES:
Time-Distance Characteristics of the Gait | up to 20 weeks
  GAITRite (CIR System INC. Clifton, NJ 07012) walkway system will be used. GAITRite; It is an electronic walkway which consists of portable carpet and sensors embedded on the carpet and transfers every foot contact to the computer when individuals walk on the carpet. With GAITRite, base of support (cm), velocity (cm / s) and cadence (steps / min) parameters will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Ali İ Yalçın, MSc, Principal Investigator — Hacettepe University; Burcu Şahin, MSc, Principal Investigator — Hacettepe University; Dilara Onan, MSc, Principal Investigator — Hacettepe University; Mert Doğan, MSc, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitation, Ankara, Altındağ, Turkey (Türkiye)